CLINICAL TRIAL: NCT01674621
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study of BA058 Administered Via a Coated Transdermal Microarray Delivery System (BA058 Transdermal) in Healthy Postmenopausal Women With Osteoporosis
Brief Title: Phase 2 Study of BA058 (Abaloparatide) Transdermal Delivery in Postmenopausal Women With Osteoporosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radius Health, Inc. (Industry)
Collaborators: Nordic Bioscience A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BA058-05-007; 2012-001921-29 (EudraCT Number)
Record Dates: First submitted 2012-08-24; First posted 2012-08-29 (Estimated); Results first posted 2016-12-19 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2020-05

CONDITIONS: Post Menopausal Osteoporosis
Keywords: BA058; Abaloparatide-SC; abaloparatide; Abaloparatide-TD; Osteo; Osteoporosis; Transdermal; Patch
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — abaloparatide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Since the abaloparatide injection arm was administered subcutaneously (SC), it was not possible to blind this arm of the study. Therefore, abaloparatide-SC was considered a reference drug, but the centralized BMD assessments and bone marker evaluations remained blinded to all treatment assignments.
Oversight: Data Monitoring Committee: No

ARMS (5):
- Abaloparatide Transdermal (50 mcg) (Experimental): Abaloparatide Transdermal Microneedle Patch - 50 microgram (mcg) daily applications for up to 6 months
  Interventions: Drug: Abaloparatide Transdermal (50 mcg)
- Abaloparatide Transdermal (100 mcg) (Experimental): Abaloparatide Transdermal Microneedle Patch - 100 mcg daily applications for up to 6 months
  Interventions: Drug: Abaloparatide Transdermal (100 mcg)
- Abaloparatide Transdermal (150 mcg) (Experimental): Abaloparatide Transdermal Microneedle Patch - 150 mcg daily applications for up to 6 months
  Interventions: Drug: Abaloparatide Transdermal (150 mcg)
- Abaloparatide Injection (80 mcg) (Active Comparator): Abaloparatide-SC Subcutaneous Injection - 80 mcg daily injections for up to 6 months
  Interventions: Drug: Abaloparatide Injection (80 mcg)
- Abaloparatide Transdermal Placebo (0 mcg) (Placebo Comparator): Abaloparatide Transdermal Microneedle Patch - 0 mcg daily applications for up to 6 months
  Interventions: Drug: Abaloparatide Placebo

INTERVENTIONS:
Drug: Abaloparatide Transdermal (50 mcg) — Abaloparatide Transdermal Microneedle Active Patch
  Other Names: BA058 Transdermal (50 mcg)
  Arms: Abaloparatide Transdermal (50 mcg)
Drug: Abaloparatide Transdermal (100 mcg) — Abaloparatide Transdermal Microneedle Active Patch
  Other Names: BA058 Transdermal (100 mcg)
  Arms: Abaloparatide Transdermal (100 mcg)
Drug: Abaloparatide Transdermal (150 mcg) — Abaloparatide Transdermal Microneedle Active Patch
  Other Names: BA058 Transdermal (150 mcg)
  Arms: Abaloparatide Transdermal (150 mcg)
Drug: Abaloparatide Injection (80 mcg) — Abaloparatide Subcutaneous Injection
  Other Names: BA058 Injection (80 mcg)
  Arms: Abaloparatide Injection (80 mcg)
Drug: Abaloparatide Placebo — Abaloparatide Transdermal Microneedle Placebo Patch
  Other Names: BA058 Placebo
  Arms: Abaloparatide Transdermal Placebo (0 mcg)

SUMMARY:
To determine the clinical safety and efficacy of abaloparatide transdermal in otherwise healthy postmenopausal women with osteoporosis as assessed by changes in bone mineral density (BMD) and serum markers of bone metabolism when compared to transdermal placebo and abaloparatide injection for 6 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal woman, less than 85 years old.
* BMD T-score ≤-2.5 of spine or hip (femoral neck) or ≤-2.0 with previous fracture (within 5 years).
* Normal physical exam, vital signs, electrocardiogram (ECG), and medical history.
* Laboratory tests within the normal range, including serum calcium, Vitamin D, parathyroid hormone (PTH) (1-84), serum phosphorus, and alkaline phosphatase.

Exclusion Criteria:

* BMD T-score ≤-5.0 at the lumbar spine or hip.
* History of bone disorders (for example, Paget's disease) other than postmenopausal osteoporosis.
* Significantly impaired renal function.
* History of any cancer.

Max Age: 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2012-09-25 (Actual); Primary Completion 2013-08-02 (Actual); Study Completion 2013-08-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (3):
  - Lakewood, Colorado
  - Atlanta, Georgia
  - Bethesda, Maryland
- Denmark (3):
  - Aalborg
  - Ballerup Municipality
  - Vejle
- Tallinn, Estonia
- Poland (2):
  - Lodz
  - Warsaw

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Abaloparatide Injection (80 mcg): Abaloparatide-Subcutaneous (SC) Injection - 80 mcg daily injections for up to 6 months
Period: Overall Study
Arm/Group | Abaloparatide Transdermal (50 mcg) | Abaloparatide Transdermal (100 mcg) | Abaloparatide Transdermal (150 mcg) | Abaloparatide Injection (80 mcg) | Abaloparatide Transdermal Placebo (0 mcg)
Started | 50 | 51 | 48 | 51 | 50
Modified Intent-to-Treat Population (Randomized participants with pretreatment and end-of-treatment evaluable radiologic assessments.) | 47 | 46 | 43 | 49 | 46
Safety Population (All participants who received 1 or more doses of study medication.) | 50 | 51 | 47 | 51 | 50
Completed | 45 | 43 | 41 | 45 | 44
Not Completed | 5 | 8 | 7 | 6 | 6
Not completed — Adverse Event | 3 | 2 | 5 | 5 | 1
Not completed — Inability to Complete Study Procedures | 0 | 0 | 0 | 0 | 2
Not completed — Severe Abaloparatide-SC Hypersensitivity | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 5 | 2 | 0 | 1
Not completed — Other than specified | 0 | 1 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat (mITT) population included randomized participants with pretreatment and end-of-treatment evaluable radiologic assessments.
Groups:
- Abaloparatide Transdermal (50 mcg): Abaloparatide Transdermal Microneedle Patch - 50 mcg daily applications for up to 6 months
- Total: Total of all reporting groups
Arm/Group | Abaloparatide Transdermal (50 mcg) | Abaloparatide Transdermal (100 mcg) | Abaloparatide Transdermal (150 mcg) | Abaloparatide Injection (80 mcg) | Abaloparatide Transdermal Placebo (0 mcg) | Total
Number analyzed (Participants) | 47 | 46 | 43 | 49 | 46 | 231
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (4.83) | 65.7 (5.26) | 66.3 (6.46) | 66.4 (5.48) | 66.5 (7.27) | 66.2 (5.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 46 | 43 | 49 | 46 | 231
  Male | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Bone Mineral Density (BMD) of Lumbar Spine at 6 Months
Description: Percent change in BMD as specified by dual energy x-ray absorptiometry (DXA) scans of the lumbar spine.
Time Frame: Baseline, 6 Months
Population: mITT population included all participants with pretreatment and end-of-treatment evaluable radiologic assessments. The participants were analyzed as randomized.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Abaloparatide Transdermal (50 mcg) | Abaloparatide Transdermal (100 mcg) | Abaloparatide Transdermal (150 mcg) | Abaloparatide Injection (80 mcg) | Abaloparatide Transdermal Placebo (0 mcg)
Number analyzed (Participants) | 47 | 46 | 43 | 49 | 46
Percent change | 1.87 (2.87) | 2.33 (2.96) | 2.95 (3.13) | 5.80 (4.21) | 0.04 (2.47)
Statistical Analysis 1: Comparison: Abaloparatide Transdermal (50 mcg) vs Abaloparatide Transdermal Placebo (0 mcg); Test type: Superiority or Other; p = 0.0066, Dunnett's test — Threshold for significance at 0.05 level; P-value from Dunnett's test comparing percent change of BMD from baseline to end-of-treatment to each transdermal dose group versus placebo
Statistical Analysis 2: Comparison: Abaloparatide Transdermal (100 mcg) vs Abaloparatide Transdermal Placebo (0 mcg); Test type: Superiority or Other; p = 0.0005, Dunnett's test — Threshold for significance at 0.05 level; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Abaloparatide Transdermal (150 mcg) vs Abaloparatide Transdermal Placebo (0 mcg); Test type: Superiority or Other; p < 0.0001, Dunnett's test — Threshold for significance at 0.05 level; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Abaloparatide Transdermal (50 mcg) vs Abaloparatide Injection (80 mcg); Test type: Superiority or Other; Mean Difference (Final Values) = -3.930, 95% CI 2-sided [-5.555 to -2.305] — Mean difference of percent change of BMD from baseline to end-of-treatment between treatment groups (transdermal and SC injection)
Statistical Analysis 5: Comparison: Abaloparatide Transdermal (100 mcg) vs Abaloparatide Injection (80 mcg); Test type: Superiority or Other; Mean Difference (Final Values) = -3.470, 95% CI 2-sided [-5.104 to -1.837] — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 6: Comparison: Abaloparatide Transdermal (150 mcg) vs Abaloparatide Injection (80 mcg); Test type: Superiority or Other; Mean Difference (Final Values) = -2.856, 95% CI 2-sided [-4.519 to -1.193] — [estimate comment as in outcome 1, analysis 4]

2. Secondary Outcome: Percent Change From Baseline in BMD of Total Hip at 6 Months
Description: Percent change in BMD as specified by DXA scans of the total hip.
Time Frame: Baseline, 6 Months
Population: mITT population included all participants with pre-treatment and end-of-treatment evaluable radiologic assessments. The participants were analyzed as randomized.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Abaloparatide Transdermal (50 mcg) | Abaloparatide Transdermal (100 mcg) | Abaloparatide Transdermal (150 mcg) | Abaloparatide Injection (80 mcg) | Abaloparatide Transdermal Placebo (0 mcg)
Number analyzed (Participants) | 47 | 46 | 43 | 49 | 46
Percent change | 0.97 (1.95) | 1.32 (1.96) | 1.49 (1.73) | 2.74 (3.05) | -0.02 (2.39)
Statistical Analysis 1: Comparison: Abaloparatide Transdermal (50 mcg) vs Abaloparatide Transdermal Placebo (0 mcg); Test type: Superiority or Other; p = 0.0547, Dunnett's test — Threshold for significance at 0.05 level; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Abaloparatide Transdermal (100 mcg) vs Abaloparatide Transdermal Placebo (0 mcg); Test type: Superiority or Other; p = 0.0056, Dunnett's test — Threshold for significance at 0.05 level; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Abaloparatide Transdermal (150 mcg) vs Abaloparatide Transdermal Placebo (0 mcg); Test type: Superiority or Other; p = 0.0018, Dunnett's test — Threshold for significance at 0.05 level; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Abaloparatide Transdermal (50 mcg) vs Abaloparatide Injection (80 mcg); Test type: Superiority or Other; Mean Difference (Final Values) = -1.768, 95% CI 2-sided [-2.864 to -0.672] — Mean difference of percent change off BMD from baseline to end-of-treatment between active treatment groups (transdermal and SC injection)
Statistical Analysis 5: Comparison: Abaloparatide Transdermal (100 mcg) vs Abaloparatide Injection (80 mcg); Test type: Superiority or Other; Mean Difference (Final Values) = -1.420, 95% CI 2-sided [-2.522 to -0.318] — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 6: Comparison: Abaloparatide Transdermal (150 mcg) vs Abaloparatide Injection (80 mcg); Test type: Superiority or Other; Mean Difference (Final Values) = -1.247, 95% CI 2-sided [-2.368 to -0.126] — [estimate comment as in outcome 1, analysis 4]

3. Secondary Outcome: Percent Change From Baseline in BMD of Forearm at 6 Months
Description: Percent change in BMD as specified by DXA scans of the forearm.
Time Frame: Baseline, 6 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Abaloparatide Transdermal (50 mcg) | Abaloparatide Transdermal (100 mcg) | Abaloparatide Transdermal (150 mcg) | Abaloparatide Injection (80 mcg) | Abaloparatide Transdermal Placebo (0 mcg)
Number analyzed (Participants) | 47 | 46 | 43 | 49 | 46
Percent change | -0.24 (2.74) | -0.16 (3.71) | 0.84 (2.96) | 0.33 (3.41) | 0.05 (3.18)
Statistical Analysis 1: Comparison: Abaloparatide Transdermal (50 mcg) vs Abaloparatide Transdermal Placebo (0 mcg); Test type: Superiority or Other; p = 0.9493, Dunnett's test — Threshold for significance at 0.05 level; P-value from Dunnett's test comparing percent change of BMD from baseline to end-of treatment to each transdermal dose group versus placebo
Statistical Analysis 2: Comparison: Abaloparatide Transdermal (100 mcg) vs Abaloparatide Transdermal Placebo (0 mcg); Test type: Superiority or Other; p = 0.9806, Dunnett's test — Threshold for significance at 0.05 level; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Abaloparatide Transdermal (150 mcg) vs Abaloparatide Transdermal Placebo (0 mcg); Test type: Superiority or Other; p = 0.5191, Dunnett's test — Threshold for significance at 0.05 level; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Abaloparatide Transdermal (50 mcg) vs Abaloparatide Injection (80 mcg); Test type: Superiority or Other; Mean Difference (Final Values) = -0.564, 95% CI 2-sided [-2.168 to 1.040] — [estimate comment as in outcome 2, analysis 4]
Statistical Analysis 5: Comparison: Abaloparatide Transdermal (100 mcg) vs Abaloparatide Injection (80 mcg); Test type: Superiority or Other; Mean Difference (Final Values) = -0.483, 95% CI 2-sided [-2.115 to 1.150] — [estimate comment as in outcome 2, analysis 4]
Statistical Analysis 6: Comparison: Abaloparatide Transdermal (150 mcg) vs Abaloparatide Injection (80 mcg); Test type: Superiority or Other; Mean Difference (Final Values) = 0.517, 95% CI 2-sided [-1.106 to 2.139] — [estimate comment as in outcome 2, analysis 4]

4. Secondary Outcome: Percent Change From Baseline in Serum Bone-Specific Alkaline Phosphatase (BSAP) at 6 Months
Time Frame: Baseline, 6 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Abaloparatide Transdermal (50 mcg) | Abaloparatide Transdermal (100 mcg) | Abaloparatide Transdermal (150 mcg) | Abaloparatide Injection (80 mcg) | Abaloparatide Transdermal Placebo (0 mcg)
Number analyzed (Participants) | 47 | 46 | 43 | 49 | 46
Percent change | -4.84 (23.87) | 5.22 (43.66) | -5.52 (37.86) | 17.30 (42.76) | 10.23 (64.93)
Statistical Analysis 1: Comparison: Abaloparatide Transdermal (50 mcg) vs Abaloparatide Transdermal Placebo (0 mcg); Test type: Superiority or Other; p = 0.2549, Dunnett's test — Threshold for significance at 0.05 level; P-value from Dunnett's test comparing percent change of BSAP from baseline to end-of-treatment to each transdermal dose group versus placebo
Statistical Analysis 2: Comparison: Abaloparatide Transdermal (100 mcg) vs Abaloparatide Transdermal Placebo (0 mcg); Test type: Superiority or Other; p = 0.9115, Dunnett's test — Threshold for significance at 0.05 level; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Abaloparatide Transdermal (150 mcg) vs Abaloparatide Transdermal Placebo (0 mcg); Test type: Superiority or Other; p = 0.2390, Dunnett's test — Threshold for significance at 0.05 level; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Abaloparatide Transdermal (50 mcg) vs Abaloparatide Injection (80 mcg); Test type: Superiority or Other; Mean Difference (Final Values) = -22.146, 95% CI 2-sided [-40.501 to -3.790] — Mean difference of percent change from baseline to end-of-treatment between active treatment groups (transdermal and SC injection)
Statistical Analysis 5: Comparison: Abaloparatide Transdermal (100 mcg) vs Abaloparatide Injection (80 mcg); Test type: Superiority or Other; Mean Difference (Final Values) = -12.086, 95% CI 2-sided [-30.543 to 6.372] — [estimate comment as in outcome 4, analysis 4]
Statistical Analysis 6: Comparison: Abaloparatide Transdermal (150 mcg) vs Abaloparatide Injection (80 mcg); Test type: Superiority or Other; Mean Difference (Final Values) = -22.828, 95% CI 2-sided [-41.614 to -4.041] — [estimate comment as in outcome 4, analysis 4]

5. Secondary Outcome: Percent Change From Baseline in Serum Procollagen Type I C Propeptide (PICP) at 6 Months
Time Frame: Baseline, 6 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Abaloparatide Transdermal (50 mcg) | Abaloparatide Transdermal (100 mcg) | Abaloparatide Transdermal (150 mcg) | Abaloparatide Injection (80 mcg) | Abaloparatide Transdermal Placebo (0 mcg)
Number analyzed (Participants) | 47 | 46 | 43 | 49 | 46
Percent change | -17.26 (22.86) | -8.42 (29.51) | -16.63 (25.11) | 10.28 (72.31) | -6.76 (31.35)
Statistical Analysis 1: Comparison: Abaloparatide Transdermal (50 mcg) vs Abaloparatide Transdermal Placebo (0 mcg); Test type: Superiority or Other; p = 0.1632, Dunnett's test — Threshold for significance at 0.05 level; P-value from Dunnett's test comparing percent change of PICP from baseline to end-of-treatment to each transdermal dose group versus placebo
Statistical Analysis 2: Comparison: Abaloparatide Transdermal (100 mcg) vs Abaloparatide Transdermal Placebo (0 mcg); Test type: Superiority or Other; p = 0.9834, Dunnett's test — Threshold for significance at 0.05 level; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Abaloparatide Transdermal (150 mcg) vs Abaloparatide Transdermal Placebo (0 mcg); Test type: Superiority or Other; p = 0.2179, Dunnett's test — Threshold for significance at 0.05 level; P-value from Dunnett's test comparing percent change of PICP from baseline to end-of-treatment (EOT) to each transdermal dose group versus placebo
Statistical Analysis 4: Comparison: Abaloparatide Transdermal (50 mcg) vs Abaloparatide Injection (80 mcg); Test type: Superiority or Other; Mean Difference (Final Values) = -27.541, 95% CI 2-sided [-48.557 to -6.525] — Mean difference of percent change from baseline to end of treatment between the active treatment groups (transdermal and SC injection)
Statistical Analysis 5: Comparison: Abaloparatide Transdermal (100 mcg) vs Abaloparatide Injection (80 mcg); Test type: Superiority or Other; Mean Difference (Final Values) = -18.702, 95% CI 2-sided [-39.835 to 2.430] — [estimate comment as in outcome 5, analysis 4]
Statistical Analysis 6: Comparison: Abaloparatide Transdermal (150 mcg) vs Abaloparatide Injection (80 mcg); Test type: Superiority or Other; Mean Difference (Final Values) = -26.914, 95% CI 2-sided [-48.424 to -5.405] — [estimate comment as in outcome 5, analysis 4]

6. Secondary Outcome: Percent Change From Baseline in Serum Osteocalcin at 6 Months
Time Frame: Baseline, 6 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Abaloparatide Transdermal (50 mcg) | Abaloparatide Transdermal (100 mcg) | Abaloparatide Transdermal (150 mcg) | Abaloparatide Injection (80 mcg) | Abaloparatide Transdermal Placebo (0 mcg)
Number analyzed (Participants) | 47 | 46 | 43 | 49 | 46
Percent change | -4.37 (19.36) | 6.67 (33.38) | -3.83 (22.01) | 69.54 (81.79) | -4.21 (27.55)
Statistical Analysis 1: Comparison: Abaloparatide Transdermal (50 mcg) vs Abaloparatide Transdermal Placebo (0 mcg); Test type: Superiority or Other; p = 1.0000, Dunnett's test — Threshold for significance at 0.05 level; P-value from Dunnett's test comparing percent change of serum osteocalcin from baseline to EOT to each transdermal dose group versus placebo
Statistical Analysis 2: Comparison: Abaloparatide Transdermal (100 mcg) vs Abaloparatide Transdermal Placebo (0 mcg); Test type: Superiority or Other; p = 0.1200, Dunnett's test — Threshold for significance at 0.05 level; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Abaloparatide Transdermal (150 mcg) vs Abaloparatide Transdermal Placebo (0 mcg); Test type: Superiority or Other; p = 0.9998, Dunnett's test — Threshold for significance at 0.05 level; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Abaloparatide Transdermal (50 mcg) vs Abaloparatide Injection (80 mcg); Test type: Superiority or Other; Mean Difference (Final Values) = -73.906, 95% CI 2-sided [-96.926 to -50.886] — [estimate comment as in outcome 5, analysis 4]
Statistical Analysis 5: Comparison: Abaloparatide Transdermal (100 mcg) vs Abaloparatide Injection (80 mcg); Test type: Superiority or Other; Mean Difference (Final Values) = -62.872, 95% CI 2-sided [-86.019 to -39.725] — [estimate comment as in outcome 5, analysis 4]
Statistical Analysis 6: Comparison: Abaloparatide Transdermal (150 mcg) vs Abaloparatide Injection (80 mcg); Test type: Superiority or Other; Mean Difference (Final Values) = -73.367, 95% CI 2-sided [-96.927 to -49.807] — [estimate comment as in outcome 5, analysis 4]

7. Secondary Outcome: Percent Change From Baseline in Serum Procollagen Type I N Propeptide (PINP) at 6 Months
Time Frame: Baseline, 6 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Abaloparatide Transdermal (50 mcg) | Abaloparatide Transdermal (100 mcg) | Abaloparatide Transdermal (150 mcg) | Abaloparatide Injection (80 mcg) | Abaloparatide Transdermal Placebo (0 mcg)
Number analyzed (Participants) | 47 | 46 | 43 | 49 | 46
Percent change | -12.76 (26.81) | 1.52 (57.29) | -6.78 (38.91) | 97.64 (172.52) | -7.26 (35.49)
Statistical Analysis 1: Comparison: Abaloparatide Transdermal (50 mcg) vs Abaloparatide Transdermal Placebo (0 mcg); Test type: Superiority or Other; p = 0.8569, Dunnett's test — Threshold for significance at 0.05 level; P-value from Dunnett's test comparing percent change of PINP from baseline to end-of-treatment to each transdermal dose group versus placebo
Statistical Analysis 2: Comparison: Abaloparatide Transdermal (100 mcg) vs Abaloparatide Transdermal Placebo (0 mcg); Test type: Superiority or Other; p = 0.6091, Dunnett's test — Threshold for significance at 0.05 level; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: Abaloparatide Transdermal (150 mcg) vs Abaloparatide Transdermal Placebo (0 mcg); Test type: Superiority or Other; p = 0.9999, Dunnett's test — Threshold for significance at 0.05 level; P-value from Dunnett's test comparing percent change of PINP from baseline to EOT to each transdermal dose group versus placebo
Statistical Analysis 4: Comparison: Abaloparatide Transdermal (50 mcg) vs Abaloparatide Injection (80 mcg); Test type: Superiority or Other; Mean Difference (Final Values) = -110.398, 95% CI 2-sided [-156.966 to -63.831] — [estimate comment as in outcome 5, analysis 4]
Statistical Analysis 5: Comparison: Abaloparatide Transdermal (100 mcg) vs Abaloparatide Injection (80 mcg); Test type: Superiority or Other; Mean Difference (Final Values) = -96.115, 95% CI 2-sided [-142.940 to -49.290] — [estimate comment as in outcome 5, analysis 4]
Statistical Analysis 6: Comparison: Abaloparatide Transdermal (150 mcg) vs Abaloparatide Injection (80 mcg); Test type: Superiority or Other; Mean Difference (Final Values) = -104.418, 95% CI 2-sided [-152.079 to -56.758] — [estimate comment as in outcome 5, analysis 4]

8. Secondary Outcome: Percent Change From Baseline in Serum Carboxy-terminal Cross-linking Telopeptide of Type I Collagen (CTXI) at 6 Months
Time Frame: Baseline, 6 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Abaloparatide Transdermal (50 mcg) | Abaloparatide Transdermal (100 mcg) | Abaloparatide Transdermal (150 mcg) | Abaloparatide Injection (80 mcg) | Abaloparatide Transdermal Placebo (0 mcg)
Number analyzed (Participants) | 47 | 46 | 43 | 49 | 46
Percent change | -2.61 (28.77) | 1.65 (48.66) | -8.22 (54.84) | 41.11 (104.12) | 9.42 (22.57)
Statistical Analysis 1: Comparison: Abaloparatide Transdermal (50 mcg) vs Abaloparatide Transdermal Placebo (0 mcg); Test type: Superiority or Other; p = 0.3483, Dunnett's test — Threshold for significance at 0.05 level; P-value from Dunnett's test comparing percent change of CTXI from baseline to end-of-treatment to each transdermal dose group versus placebo
Statistical Analysis 2: Comparison: Abaloparatide Transdermal (100 mcg) vs Abaloparatide Transdermal Placebo (0 mcg); Test type: Superiority or Other; p = 0.6839, Dunnett's test — Threshold for significance at 0.05 level; [statistical method as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Abaloparatide Transdermal (150 mcg) vs Abaloparatide Transdermal Placebo (0 mcg); Test type: Superiority or Other; p = 0.1067, Dunnett's test — Threshold for significance at 0.05 level; [statistical method as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Abaloparatide Transdermal (50 mcg) vs Abaloparatide Injection (80 mcg); Test type: Superiority or Other; Mean Difference (Final Values) = -43.721, 95% CI 2-sided [-75.748 to -11.694] — [estimate comment as in outcome 5, analysis 4]
Statistical Analysis 5: Comparison: Abaloparatide Transdermal (100 mcg) vs Abaloparatide Injection (80 mcg); Test type: Superiority or Other; Mean Difference (Final Values) = -39.461, 95% CI 2-sided [-71.665 to -7.257] — [estimate comment as in outcome 5, analysis 4]
Statistical Analysis 6: Comparison: Abaloparatide Transdermal (150 mcg) vs Abaloparatide Injection (80 mcg); Test type: Superiority or Other; Mean Difference (Final Values) = -49.334, 95% CI 2-sided [-82.113 to -16.555] — [estimate comment as in outcome 5, analysis 4]

9. Secondary Outcome: Number of Participants With Abnormal Physical Examinations at Screening and End of Treatment (6 Months)
Description: A full physical examination included, at a minimum: general appearance, skin, head/ears/eyes/nose/throat, lungs/chest, breasts, heart, abdomen, lymph nodes, musculoskeletal, extremities, and neurologic. Physical examination results that were considered abnormal were determined by the Investigator. A summary of other non-serious adverse events (AEs) and all serious AEs (SAEs), regardless of causality is located in Reported AE section.
Time Frame: Baseline up to 6 Months
Population: Safety population included all participants who received 1 or more doses of study medication. The participants were analyzed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Abaloparatide Transdermal (50 mcg) | Abaloparatide Transdermal (100 mcg) | Abaloparatide Transdermal (150 mcg) | Abaloparatide Injection (80 mcg) | Abaloparatide Transdermal Placebo (0 mcg)
Number analyzed (Participants) | 50 | 51 | 47 | 51 | 50
Participants
  General appearance at Screening | 0 | 0 | 0 | 1 | 0
  General appearance at 6 months | 0 | 0 | 1 | 1 | 0
  Skin at Screening | 28 | 24 | 17 | 14 | 21
  Skin at 6 months | 29 | 26 | 16 | 14 | 17
  Head at Screening | 6 | 3 | 2 | 5 | 1
  Head at 6 months | 6 | 4 | 3 | 4 | 2
  Lungs at Screening | 0 | 0 | 0 | 1 | 1
  Lungs at 6 months | 0 | 0 | 0 | 1 | 0
  Breasts at Screening | 4 | 7 | 3 | 3 | 11
  Breasts at 6 months | 4 | 7 | 3 | 4 | 10
  Abdomen at Screening | 7 | 8 | 4 | 9 | 4
  Abdomen at 6 months | 6 | 7 | 3 | 9 | 3
  Lymph nodes at Screening | 0 | 0 | 1 | 0 | 0
  Lymph nodes at 6 months | 0 | 0 | 0 | 0 | 1
  Columna at Screening | 1 | 3 | 7 | 4 | 1
  Columna at 6 months | 1 | 2 | 7 | 3 | 1
  Extremities at Screening | 21 | 13 | 14 | 23 | 21
  Extremities at 6 months | 23 | 10 | 14 | 25 | 21
  Neurologic at Screening | 0 | 0 | 0 | 2 | 1
  Neurologic at 6 months | 0 | 0 | 0 | 3 | 1

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) That Occurred During the Study That Were Associated With Vital Sign Changes
Description: Vital sign parameters included respiration rate (breaths/minute), body temperature (°C), systolic blood pressure (SBP) and diastolic blood pressure (DBP) (mmHg), and heart rate (bpm). Number of participants for each TEAE is presented. The same participant may be included in more than one TEAE category. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to 7 Months
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Abaloparatide Transdermal (50 mcg) | Abaloparatide Transdermal (100 mcg) | Abaloparatide Transdermal (150 mcg) | Abaloparatide Injection (80 mcg) | Abaloparatide Transdermal Placebo (0 mcg)
Number analyzed (Participants) | 50 | 51 | 47 | 51 | 50
Participants
  Hypertension | 0 | 1 | 0 | 0 | 0
  Blood Pressure Increased | 0 | 0 | 1 | 1 | 0
  Heart Rate increased | 0 | 0 | 1 | 0 | 0
  Dyspnoea | 0 | 0 | 0 | 1 | 0
  Dizziness | 0 | 0 | 0 | 1 | 0

11. Secondary Outcome: Number of Participants With a Clinically Meaningful Abnormal Electrocardiogram (ECG) Test Result
Description: The following ECG parameters were recorded: rhythm, heart rate, PR interval, QRS duration and QT/QTc. ECG results that were considered clinically meaningful were to be determined by the Investigator. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to 7 Months
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Abaloparatide Transdermal (50 mcg) | Abaloparatide Transdermal (100 mcg) | Abaloparatide Transdermal (150 mcg) | Abaloparatide Injection (80 mcg) | Abaloparatide Transdermal Placebo (0 mcg)
Number analyzed (Participants) | 50 | 51 | 47 | 51 | 50
Participants | 0 | 0 | 1 | 2 | 0

12. Secondary Outcome: Number of Participants With an Abnormal Clinical Hematology Laboratory Parameter With an Eastern Cooperative Oncology Group (ECOG) Score of Grade 3 or Grade 4
Description: Hematology laboratory parameters that were evaluated via ECOG Grade 3 and Grade 4 criteria (presented in parentheses) included: white blood cell (Grade 3: 1.0-1.9*10^9/liter [L]; Grade 4 <1.0*10^9/L), platelets (Grade 3: 25.0-49.9*10^9/L; Grade 4: <25.0*10^9/L), haemoglobin (Grade 3: 65.0-79.0 grams [g]/L or 4.0-4.9 mmol/L; Grade 4: <65.0 g/L or <4.0 millimole [mmol]/L), granulocytes/bands (Grade 3: 0.5-0.9*10^9/L; Grade 4: <0.5*10^9/L), lymphocytes (Grade 3: 0.5-0.9*10^9/L; Grade 4: <0.5 *10^9/L), haemorrhage (Grade 3: gross, 3 - 4 units transfusion per episode; Grade 4: massive, > 4 units transfusion per episode). A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to 6 Months
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Abaloparatide Transdermal (50 mcg) | Abaloparatide Transdermal (100 mcg) | Abaloparatide Transdermal (150 mcg) | Abaloparatide Injection (80 mcg) | Abaloparatide Transdermal Placebo (0 mcg)
Number analyzed (Participants) | 50 | 51 | 47 | 51 | 50
Participants | 6 | 5 | 4 | 1 | 5

13. Secondary Outcome: Number of Participants With an Abnormal Clinical Chemistry Laboratory Parameter With an ECOG Score of Grade 3 or Grade 4
Description: Chemistry laboratory parameters that were evaluated via ECOG Grade 3 and Grade 4 criteria (presented in parentheses) included: sodium, potassium, chloride, inorganic phosphorus, albumin, total protein (Grade 3: 4 (+), >1.0 g%, or >10 g/L; Grade 4: nephrotic syndrome), glucose, blood urea nitrogen (BUN), creatinine (Grade 3: 3.1-6.0*normal; Grade 4: >6.0*normal), uric acid, aspartate aminotransferase (AST) (Grade 3: 5.1-20.0 units [U]/L*normal, Grade 4: >20.0 U/L*normal), alanine aminotransferase (ALT) (Grade 3: 5.1-20.0 U/L*normal; Grade 4: >20.0 U/L*normal), gamma-glutamyltranspeptidase (GGT), creatine phosphokinase (CPK), alkaline phosphatase (Grade 3: 5.1-20.0 U/L*normal; Grade 4: >20.0 U/L*normal), total bilirubin (Grade 3: 1.5-3.0*normal; Grade 4: >3.0*normal), lactate dehydrogenase (LDH), cholesterol, triglycerides, total calcium. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to 6 Months
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Abaloparatide Transdermal (50 mcg) | Abaloparatide Transdermal (100 mcg) | Abaloparatide Transdermal (150 mcg) | Abaloparatide Injection (80 mcg) | Abaloparatide Transdermal Placebo (0 mcg)
Number analyzed (Participants) | 50 | 51 | 47 | 51 | 50
Participants | 1 | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With an Abnormal Clinical Coagulation Laboratory Parameter With an ECOG Score of Grade 3 or Grade 4
Description: Coagulation laboratory parameters that were evaluated via ECOG Grade 3 and Grade 4 criteria (presented in parentheses) included: prothrombin time (quick) (Grade 3: 1.51%-2.00%*normal, Grade 4: >2.00%*normal), partial thromboplastin time (Grade 3: 2.34-3.00 seconds [sec], Grade 4: >3.00 secs*normal). A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to 6 Months
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Abaloparatide Transdermal (50 mcg) | Abaloparatide Transdermal (100 mcg) | Abaloparatide Transdermal (150 mcg) | Abaloparatide Injection (80 mcg) | Abaloparatide Transdermal Placebo (0 mcg)
Number analyzed (Participants) | 50 | 51 | 47 | 51 | 50
Participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 7 Months
Description: Safety population included all participants who received 1 or more doses of study medication. The participants were analyzed as treated.
Arm/Group | Abaloparatide Transdermal (50 mcg) | Abaloparatide Transdermal (100 mcg) | Abaloparatide Transdermal (150 mcg) | Abaloparatide Injection (80 mcg) | Abaloparatide Transdermal Placebo (0 mcg)
Serious Adverse Events (participants affected / at risk) | 0/50 | 2/51 | 2/47 | 4/51 | 1/50
Other Adverse Events (participants affected / at risk) | 40/50 | 40/51 | 37/47 | 41/51 | 39/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abaloparatide Transdermal (50 mcg) (N=50) | Abaloparatide Transdermal (100 mcg) (N=51) | Abaloparatide Transdermal (150 mcg) (N=47) | Abaloparatide Injection (80 mcg) (N=51) | Abaloparatide Transdermal Placebo (0 mcg) (N=50)
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abaloparatide Transdermal (50 mcg) (N=50) | Abaloparatide Transdermal (100 mcg) (N=51) | Abaloparatide Transdermal (150 mcg) (N=47) | Abaloparatide Injection (80 mcg) (N=51) | Abaloparatide Transdermal Placebo (0 mcg) (N=50)
Palpitations (Cardiac disorders) | 0 | 2 | 0 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 3 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 6 | 3 | 2
Application site erythema (General disorders) | 4 | 5 | 4 | 0 | 2
Application site pruritus (General disorders) | 0 | 1 | 4 | 0 | 0
Influenza like illness (General disorders) | 1 | 3 | 1 | 1 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 4 | 1 | 1
Cystitis (Infections and infestations) | 2 | 0 | 4 | 1 | 1
Influenza (Infections and infestations) | 4 | 4 | 2 | 5 | 4
Nasopharyngitis (Infections and infestations) | 11 | 10 | 8 | 13 | 9
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 3 | 1 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 3 | 3 | 5
Dizziness (Nervous system disorders) | 2 | 2 | 3 | 8 | 1
Headache (Nervous system disorders) | 2 | 2 | 5 | 5 | 5
Hypercalciuria (Renal and urinary disorders) | 0 | 1 | 2 | 3 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3 | 0 | 1
Injection site erythema (General disorders) | 0 | 0 | 0 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results may not be published prior to the Study Report completion. Investigators may publish results, providing a manuscript to the Sponsor =/> 30 days prior to its submission to a publisher. Sponsor will provide manuscript to Investigators =/> 30 days prior to its submission. Investigator shall comply with Sponsor's policy, withholding publication for an additional 60 days to permit the Sponsor to obtain patent or other proprietary rights protection, if deemed necessary.